CLINICAL TRIAL: NCT00587886
Title: Estrogen, Diet, Genetics and Endometrial Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other); Municipal Institute of Medical Research (Unknown); Department of Health and Human Services (U.S. Federal Agency); Penn State University (Other)
Responsible Party: Sponsor
Other Study IDs: 01-119; CA83918
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Endometrial Cancer; Ovarian Cancer; Corpus Uteri; Endometrium
Keywords: Cancer; Endometrial cancer; Ovarian cancer; Corpus Uteri; Endometrium
MeSH Terms: conditions — Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal specimen

GROUPS / COHORTS (2):
- Cases: Cases will be women with newly diagnosed endometrial or ovarian cancer who are residents of six counties in New Jersey.
  Interventions: Behavioral: Questionnaire
- Controls: Controls will be selected from the general population in those counties by use of random digit dialing for those under 65 years of age, from Centers for Medicare and Medicaid Services (CMS) lists for those aged 65 years and over, and from neighborhood sampling.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — The main questionnaire will cover established risk and protective factors for endometrial and ovarian cancer, as well as other possible risk factors. This includes: menstrual history; pregnancy history; use of hormones for menopausal symptoms or other reasons; smoking history; height and weight; use of oral contraceptives and other methods of birth control; family history of cancer; medical history; demographic characteristics. We will also collect dietary data using the Gladys Block questionnaire, to which we have added a supplement to measure consumption of phytoestrogens. We will also obtain a buccal sample from each respondent as the source of DNA for genetic analysis.
  Groups: Cases
Behavioral: Questionnaire — The main questionnaire will cover established risk and protective factors for endometrial and ovarian cancer, as well as other possible risk factors. This includes: menstrual history; pregnancy history; use of hormones for menopausal symptoms or other reasons; smoking history; height and weight; use of oral contraceptives and other methods of birth control; family history of cancer; medical history; demographic characteristics. We will also collect dietary data using the Gladys Block questionnaire, to which we have added a supplement to measure consumption of phytoestrogens. We will also obtain a buccal sample from each respondent as the source of DNA for genetic analysis.
  We will conduct interviews mainly by telephone but also in person (at home or another convenient place)if the participant prefers.
  Groups: Controls

SUMMARY:
The purpose of this study is to see how people's diets, other aspects of their lifestyles, and their individual genetic makeup affect their chances of getting endometrial cancer (cancer of the uterus).

This survey will enroll several hundred women who have or have had endometrial cancer and several hundred who do not. We will compare these two groups of women to see what factors may lead to endometrial cancer.

DETAILED DESCRIPTION:
We will conduct a population-based case-control study in six counties of New Jersey. Cases will be women with newly-diagnosed endometrial or ovarian cancer. Controls will be matched by 5-year age groups and selected by random digit dialing (for those under 65), from Centers for Medicare and Medicaid Services (CMS) files (for those 65 and over), or from neighborhood sampling. Controls will not have had a hysterectomy.

There will be 400 cases with endometrioid tumors, 60 with serous tumors or clear cell tumors, 300 with ovarian cancer, and 400 controls. In addition, there will be a small group of black women included from MSKCC.

We will interview participants about known and potential risk factors for endometrial and ovarian cancer and obtain information on diet. We will obtain DNA for genetic analysis from buccal specimens collected using a mouthwash rinse method. We will use logistic regression to determine odds ratios for disease with various exposures. For endometrial cancer, we will examine the association of risk with genotypes in strata defined by body mass index and dietary fat consumption.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with epithelial endometrial or ovarian cancer within the year before being contacted (cases)
* Aged 21 and over
* Residents of Essex, Union, Morris, Middlesex, Bergen, or Hudson counties, NJ
* Black women with and without endometrial cancer who are seeing gynecologists at MSKCC

Exclusion Criteria:

* Unable to sign informed consent
* Consent withheld by physician (cases)
* Hysterectomy (controls)
* Do not speak English or Spanish

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In collaboration with the New Jersey Department of Health and Senior Services NJDHSS), we will use rapid case ascertainment to identify patients as they are diagnosed.For controls aged 65 and over, we will obtain lists from CMS of a sample of women in the 6 counties. As an alternative way of reaching controls, we will conduct area sampling.
Sampling Method: Probability Sample
Enrollment: 1315 (Actual)
Dates: Start 2001-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate the role of weight, diet, and individual genetic susceptibility to endometrial cancer | 3 years

SECONDARY OUTCOMES:
The secondary aim of this study is to obtain epidemiologic data on papillary serous and clear cell histologic types of endometrial cancer. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mengmeng Du, ScD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org